CLINICAL TRIAL: NCT00282789
Title: BiPAP for Cardiomyopathy With Central Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nagoya University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU-06-A-0002
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2006-01-30 (Estimated); Status verified 2000-06

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Device: bilevel positive airway pressure
Device: bilevel positive airway pressure (Device)

SUMMARY:
We investigated whether treatment of central sleep apnea-hypopnea with bilevel positive airway pressure (BiPAP) in patients with idiopathic dilated cardiomyopathy (IDCM) would improve LV function.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic dilated cardiomyopathy

Exclusion Criteria:

* a history of alcohol abuse, diabetes mellitus, endocrine disorders, hypertension, obstructive sleep apnea syndrome, and chronic obstructive pulmonary disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuhiro Yokota, MD,PhD, Study Chair — Department of Cardiovascular Genome Science, Nagoya University School of Medicine, Nagoya, Aichi, Japan
Locations (1):
- Nagoya University of Health Sciences, Nagoya, Japan